CLINICAL TRIAL: NCT02713152
Title: POSAG: Prevalence of Obstructive Sleep Apnoea in Glaucoma
Brief Title: Prevalence of Obstructive Sleep Apnoea in Glaucoma
Acronym: POSAG
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Anglia Ruskin University (Other); Hinchingbrooke Healthcare NHS Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: P02058
Record Dates: First submitted 2016-01-25; First posted 2016-03-18 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnoea; Open Angle Glaucoma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with OAG: Patients with a diagnosis of Open Angle Glaucoma
- Controls: Controls without a diagnosis of Open Angle Glaucoma

SUMMARY:
This study aims to investigate a potential link between Obstructive Sleep Apnoea (OSA) and Open Angle Glaucoma (OAG); initially by determining whether the prevalence of OSA is higher in patients with OAG in comparison to people without glaucoma and if OSA is an independent risk factor for OAG. It will comprehensively phenotype glaucoma patients for variables that may be associated with both OSA and OAG.

DETAILED DESCRIPTION:
Open Angle Glaucoma (OAG) is an eye disease which can lead to irreversible loss of vision caused by damage to the optic nerve at the back of the eye. It is often associated with raised fluid pressure in the eye and treated by lowering this pressure. However, despite treatment, some patients continue to lose vision and it is suspected that other factors are contributing to the optic nerve damage. Among them is Obstructive Sleep Apnoea (OSA), though the link between OAG and OSA is controversial.

This study aims to determine whether the prevalence of OSA is higher in patients with OAG in comparison to people without glaucoma. In addition, it will establish whether OSA is an independent risk factor for OAG and whether a future randomised controlled trial assessing the impact of OSA treatment with Continues Positive Airway Pressure (CPAP) on OAG outcomes would be acceptable and feasible in this population. The usefulness of OSA screening tools, including oximetry and questionnaires will also be determined. We comprehensively phenotype glaucoma patients using novel techniques, which include angiographic ocular coherence tomography and retinal oximetry. Ocular perfusion pressure will be calculated based on central retinal vein pressure measured by ophthalmodynamometry.

The study is a collaborative project between sleep specialists at Papworth Hospital and ophthalmologists at Hinchingbrooke Hospital and will involve patients attending glaucoma clinic and their relatives who will act as a control group. Two study visits will be required on consecutive days. Participants will undergo a comprehensive ocular examination and a sleep study in the form of respiratory polysomnography (respiratory PSG) at home. A brief medical history focused on cardiovascular and metabolic co-morbidities will be taken.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma patients:

1. Open angle glaucoma (including primary open angle glaucoma, normal tension glaucoma and pseudoexfoliation glaucoma) in either eye.
2. Age ≥18 years
3. Able to give informed consent and attend at the required frequency for the duration of the study.

Control group:

1. Age ≥18 years
2. Able to give informed consent and attend at the required frequency for the duration of the study.

Exclusion Criteria:

Glaucoma patients:

1. Unable to perform reliable visual field testing (>15% false positives, >20% fixation losses. However, if fixation losses are >20%, the eye tracker may be used to assess reliability)
2. Known or suspected pregnancy.
3. Tracheostomy
4. Use of nocturnal oxygen for indications other than sleep related breathing disorders (SBD).

Control group:

1. Known or suspected pregnancy
2. Known or suspected glaucoma (participants with glaucoma diagnosed during screening ophthalmic examination and newly identified glaucoma 'suspects' will also be excluded)
3. Inability to undergo screening ophthalmic examination
4. Tracheostomy
5. Use of nocturnal oxygen for indications other than sleep related breathing disorders (SBD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2016-03; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Diagnosis of OSA | Within 24 hours of recruitment on to study (cross-sectional)
  Clinical diagnosis of OSA defined as apnoea hypopnoea index (AHI) >5

SECONDARY OUTCOMES:
OSA severity | 24 hours
  OSA severity will be determined by Apnoea-Hypopnea Index (AHI) and nocturnal oxygen desaturation levels (recording from nocturnal oximetry), which are used to indicate the severity of obstructive sleep apnoea.
Glaucoma severity | 24 hours
  Glaucoma severity measured by mean deviation (MD) derived from visual fields examination
Ocular perfusion pressure (OPP) | 24 hours
  Ocular perfusion pressure will be calculated based on the following formula : OPP=2/3MAP-CVRP where MAP is mean arterial pressure and CVRP is central retinal venous pressure measured by ophthalmodymamometry.
Postural changes in intraocular pressure (IOP) | 24 hours
  Postural changes of IOP will be measured as the difference between IOP in the upright position and then supine position.
Optic nerve head perfusion | 24 hours
  Optic nerve head flow index will be measured non-invasively by Angiographic Ocular Coherence Tomography (aOCT)
Structural changes of the optic nerve | 24 hours
  Structural changes of the optic nerve will be characterised by retinal nerve fibre layer (RNFL) thickness measured by Ocular Coherence Tomography
Stop-Bang questionnaire as screening tool | 24 hours
  Sensitivity and specificity of Stop-Bang questionnaire in detecting OSA in OAG, using Stop-Bang questionnaire summary score.
Nocturnal oximetry as screening tool | 24 hours
  Sensitivity and specificity of nocturnal oximetry in detecting OSA in OAG
Diagnosis of obstructive sleep apnoea syndrome (OSAS) | 24 hours
  Prevalence of OSAS in OAG patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hinchingbrooke Hospital NHS Foundation Trust, Huntingdon, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will not be sharing individual participant data. All study data will be anonymised.